CLINICAL TRIAL: NCT00464542
Title: Asymptomatic Bacterial Vaginosis and Herpes Simplex Virus Type 2 Shedding
Brief Title: Asymptomatic Bacterial Vaginosis and Herpes Simplex Virus Type 2 (BV/HSV-2) Shedding Study
Acronym: MASH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO07030124
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-04

CONDITIONS: Bacterial Vaginosis
Keywords: herpes simplex virus
MeSH Terms: conditions — Vaginosis, Bacterial; Herpes Simplex | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metronidazole (Other): Observational before and after treatment Drug: Metronidazole 500 mg, taken by mouth, two times a day, 7 days
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — 500 mg, taken by mouth, two times a day, 7 days
  Other Names: Flagyl

SUMMARY:
This investigation assessed the effects of asymptomatic BV on daily genital tract shedding of HSV-2 by determining shedding frequency before and after treatment of asymptomatic BV.

DETAILED DESCRIPTION:
An important contributor to the epidemic spread of herpes simplex virus type 2 (HSV-2) is its high frequency of asymptomatic shedding in the genital tract, as transmission usually occurs during these periods of subclinical reactivation of the virus. Therefore, an improved understanding of the risk factors associated with HSV-2 shedding is needed.

Preliminary data suggests that bacterial vaginosis (BV) may be associated with increased genital tract shedding of HSV-2. As BV is the most common cause of vaginal symptoms in reproductive age women, even modest associations with genital tract shedding of HSV-2 would result in substantial attributable risks for transmission of the virus.

This study assessed the effects of asymptomatic BV on daily genital tract shedding of HSV-2 by determining shedding frequency before and after treatment of asymptomatic BV. Twelve HSV-2 seropositive women with asymptomatic BV were enrolled. These women were instructed to self-collect daily swab specimens for HSV-2 deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) analysis from the lower genital tract for one month. At the end of the one month follow-up visit, each participant completed a one week course of oral metronidazole for treatment of BV. This was followed by daily home collection of genital tract swab specimens for an additional one month.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-26 years old of age
* Only those women who deny symptoms of vaginal discharge and odor but who meet Amsel and Gram stain criteria for the diagnosis of BV will be eligible
* Amsel criteria (3 of the following 4 conditions) (10):
* Homogenous vaginal discharge
* Vaginal pH > 4.5
* Positive amine (sniff) test
* Presence of clue cells in the vaginal fluid
* Gram stain criteria (11):
* Score: 0-3; classification: normal; vaginal bacteria morphotype: Lactobacillus predominant
* Score: 4-6; classification: intermediate; vaginal bacteria morphotype: Lactobacilli reduced
* Score: 7-10; classification: BV; vaginal bacteria morphotype: Lactobacillus replaced by Gardnerella and anaerobes
* Eligible women will need to test positive for HSV-2 type-specific antibodies. Determination of HSV-2 serostatus will be determined by a point-of-care type-specific immunoassay kit.
* Patients capable of providing written informed consent
* Patients willing to refrain from the use of intravaginal products (i.e., contraceptive creams, gels, foams, sponges, lubricants, douches, etc.) during the study period
* Patients willing to refrain from the use of any systemic or topical genital antiviral medication during the study period
* Patients willing and capable of cooperating to the extent and degree required by this protocol

Exclusion Criteria:

* HSV-2 seronegativity (as determined by the point-of-care immunoassay)
* Pregnancy (all women will receive a pregnancy test prior to enrollment) or those women currently not practicing an effective method of birth control
* Current Chlamydia trachomatis, Neisseria gonorrhea, or Trichomonas vaginalis infection
* Use of prescriptive antiviral treatment for presumed HSV reactivation within the 14 days prior to enrollment
* Use of systemic antimicrobials within the past 14 days
* History of hypersensitivity or inability to tolerate systemic metronidazole therapy
* Nursing mother
* Patients with intrauterine devices
* Unwillingness to refrain from initiation of antiviral medication during study period
* Unwillingness to refrain from use of douche products during study period
* Unwillingness to refrain from the ingestion of any alcoholic beverages during the one-week course of oral metronidazole therapy

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Cherpes, Principal Investigator — Univerisity of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Magee Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve HSV-2 seropositive women with asymptomatic BV were enrolled. Two of these women were lost to follow-up within 2 weeks of enrollment. A third woman was lost to follow-up after initiating metronidazole therapy at study midpoint.
Groups:
- MASH Cohort: This cohort consisted of women who were seropositive for Herpes Simplex Virus type 2 (HSV-2)and who had asymptomatic bacterial vaginosis as assessed by Amsel's criteria at enrollment
Period: Pre-treatment
Arm/Group | MASH Cohort
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Post-treatment
Arm/Group | MASH Cohort
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MASH Cohort
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bacterial Vaginosis Recurrence
Description: Bacterial vaginosis, defined as any vaginal smear with a Nugent score of 7-10 during the 30 day period following cessation of metronidazole therapy.
Time Frame: 30 days after cessation of metronidazole therapy
Population: per protocol
Measure: Number; unit: Participants
Groups:
- Post-treatment MASH Cohort: Women who were seropositive for Herpes Simplex Virus type 2 (HSV-2)and had asymptomatic bacterial vaginosis as assessed by Amsel's criteria at enrollment and who provided daily vaginal smears for 30 days following cessation of metronidazole therapy
Arm/Group | Post-treatment MASH Cohort
Number analyzed (Participants) | 9
Participants | 8

2. Secondary Outcome: Median Time to Bacterial Vaginosis During the 30 Days After Cessation of Metronidazole Therapy
Description: The time by which half of the participants were diagnosed with bacterial vaginosis, defined as any vaginal smear with a Nugent score of 7-10 during the 30 day period following cessation of metronidazole therapy
Time Frame: 30 days after cessation of metronidazole therapy
Measure: Median (Full Range); unit: Days
Arm/Group | Post-treatment MASH Cohort
Number analyzed (Participants) | 9
Days | 14 [7 to 24]

ADVERSE EVENTS:
Arm/Group | MASH Cohort
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Inadequate controls (study would have been improved by inclusion of women without herpes simplex virus type 2 infection) to better determine the strength of the association between recalcitrance of BV and HSV-2 infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes